CLINICAL TRIAL: NCT06631599
Title: Effects of Different Trainings on Physical Performance in Amateur Soccer Players at Different Age
Brief Title: Effects of Trainings on Physical Performance in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AWF_AT_1
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Health; Sport; Soccer Performance; Soccer Training
Keywords: soccer; fitness; trainig; strength; speed
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): This group performed routine soccer training
- sprint training group (Experimental): This group performed, in addition to routine soccer training, sprint training with resistance
  Interventions: Other: Physical training
- Functional training group (Experimental): This group performed, in addition to routine football training, functional training
  Interventions: Other: Physical training

INTERVENTIONS:
Other: Physical training — The intervention consisted of physical exercise according to various protocols
  Other Names: speed training; functional training
  Arms: Functional training group; sprint training group

SUMMARY:
The main objective of study was to examine the effects of different trainings on physical performance in amateur soccer players at different age. Participants trained according to various training protocols aimed at improving their motor skills (strength, power, speed, efficiency). We searched for the most optimal protocol, i.e. one that most effectively improves the study of motor skills and fitness.

ELIGIBILITY:
Inclusion Criteria:

* healthy male soccer players
* amatour

Exclusion Criteria:

* any diseases
* injury

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
speed | after 4 weeks of training
  Sprinting performance (20 m distance) was measured using a radar technology
power | after 4 weeks of training
  Muscle power was measured during a vertical countermovement jump
force-velocity profile | after 4 weeks of training
  Individual force-velocity relationships were extrapolated from a spreadsheet of sprint acceleration force-velocity profiling

CONTACTS AND LOCATIONS:
Locations (1):
- Academy of Applied Sciences, Tarnów, Tarnow, Poland

IPD SHARING:
Plan to Share IPD: No